CLINICAL TRIAL: NCT06114732
Title: Motivating Physical Activity With Behavioural interVention and Electrical Stimulation Remotely in People With Intermittent Claudication (MAvERIC): a Feasibility Randomised Controlled Trial
Brief Title: Motivating Physical Activity With Behavioural interVention and Electrical Stimulation Remotely in Intermittent Claudication
Acronym: MAvERIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Glasgow Caledonian University (Other)
Collaborators: King's College London (Other); St George's, University of London (Other); University of Glasgow (Other); NHS Lanarkshire (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 332468; HLS/PSWAHS/22/224 (Other: HLS Ethics Committee GCU)
Record Dates: First submitted 2023-10-30; First posted 2023-11-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Peripheral Artery Disease; Intermittent Claudication
Keywords: Transcutaneous electrical nerve stimulation; Electrical Stimulation; Pain Management; Physiotherapy; Education; Motivational Interviewing; Feasibility
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication; Agnosia | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Walking exercise behaviour change intervention + TENS (Experimental): Participants in the Intervention groups will be asked to attend four telehealth appointments with a physiotherapist. They will also be provided with a TENS machine and training at the baseline appointment on how to use it. They will be instructed to use it daily as their symptoms require for 12 weeks. The device will be set at High Frequency-TENS (120 Hz, 200µs and a patient-determined intensity of ''strong but comfortable'').
  Interventions: Behavioral: Walking exercise behaviour change intervention + TENS
- Usual Care control (No Intervention): Usual Care at NHS Lanarkshire Vascular Services and/or Intermittent Claudication service.

INTERVENTIONS:
Behavioral: Walking exercise behaviour change intervention + TENS — MOSAIC: Participants in this group receive two 60-minute individual video telehealth consultations (on weeks one & two) and two 20-minute follow-up telephone calls (weeks six & 12) delivered at a convenient time over the internet. All sessions are delivered by a trained senior/band 6 physiotherapist. All participants randomized to this arm are provided with a pedometer and a patient manual which include information on intermittent claudication (IC), risk factors, walking guidelines, goal setting, problem solving and action planning worksheets and a walking diary.
  HF-TENS - TENS is a form of electrical stimulation that provides symptomatic pain relief that is used extensively within the health-care setting. It is a non-invasive modality; packaged in a small, portable unit that is easy to apply via small electrodes placed on the skin. Participants will be asked to use TENS during their everyday walking-based tasks, and any planned walking activity they undertake.
  Arms: Walking exercise behaviour change intervention + TENS

SUMMARY:
Peripheral Arterial Disease (PAD) is a common vascular disease which commonly causes limb pain and reduced exercise tolerance termed Intermittent Claudication (IC). People with PAD and IC have impaired quality of life, reduced walking ability, and increased mortality compared to those who do not have the condition.

Improving physical activity (PA) is important in individuals with IC it can improve function, morbidity and mortality rates. While supervised exercise classes are recommended by healthcare authorities they are geographically sparse, and not always accessible due to individuals walking limitations. While home-based exercise can be accessible and improve walking ability, it can be challenging for people with IC to initially plan, conduct, and stay motivated to complete a walking program unsupported, especially when they experience limb pain when walking.

Investigators have shown that Transcutaneous Electrical Nerve Stimulation (TENS), a non-invasive pain management device, with aims to improve pain and walking distances in patients with IC may be an acceptable modality alongside advice and support from a physiotherapist to overcome these challenges. Investigators have also shown that motivational interviewing, education, and goal-setting with a physiotherapist (physical therapist) has the potential to increase PA, and quality of life.

This study aims to conduct a feasibility trial of four telehealth physiotherapy sessions, alongside the provision of a CE-marked TENS device to reduce limb pain during physical activity. This will be compared to the usual care offered in NHS Lanarkshire

DETAILED DESCRIPTION:
Peripheral Arterial Disease (PAD) is a common vascular disease which is symptomatic in 2.4% of 50 to 89 year olds in the UK population. Symptomatic PAD initially presents clinically as limb pain and reduced exercise intolerance termed Intermittent Claudication (IC). Patients with PAD and IC have impaired quality of life due to reduced physical capacity and 3-4 times increased mortality compared to age and sex matched controls.

Improving daily physical activity (PA) is particularly important in individuals with IC as lower PA levels have been recognised as a strong predictor of increased morbidity and mortality in this population. Supervised exercise programs are recommended in clinical guidelines with proven efficacy to help increase physical activity, improve quality of life and contribute to secondary prevention of adverse cardiovascular events (ACVE). Despite this, provision of classes is varied geographically in the UK, and generally is centralised away from rural areas, which may limit uptake and adherence. An alternative to this exercise format may be home-based exercise in the format of a walking-based behaviour change intervention. Home-based exercise for people with intermittent claudication demonstrate a low number of related adverse events, and in the case of walking-based programmes, are likely more accessible, require little equipment, and involve increasing an activity of daily living (ADL) in people with intermittent claudication. Therefore, there is a need for investigation to the acceptability of novel methods of increasing physical activity in a home-based setting.

Lack of self-efficacy, attributed to poor understanding of the disease and uncertainty regarding the importance of exercise, has been shown to be a major barrier to exercise uptake in patients with PAD and IC. Moreover, home based exercise for the self-management of IC is less established in the literature than SEP and there are concerns of low adherence without clinician monitoring. However, if an engaging intervention feasible to the patient and healthcare provider can be established there is potential for greater equality in care, reduced healthcare utilisation and improvement of self-management of PAD in the population.

A proposed intervention to augment walking based physical activity is Transcutaneous electrical nerve stimulation (TENS). TENS a low-cost, non-invasive pain management device with aims to improve pain and walking distances in patients with IC. In our exploratory study we demonstrated that TENS applied to the lower limb during treadmill walking significantly improved pain and increased treadmill walking distances above placebo levels. In addition, Motivating Structured Walking Activity in People with Intermittent Claudication (MOSAIC) is a walking based behavioural intervention utilising motivational interviewing to help people with PAD and IC increase their physical activity. This may help patients plan and overcome barriers to increasing their physical activity by joint clinician and patient set physical activity goals. Both TENS and MOSAIC have potential for remote delivery which could have effects on secondary prevention of ACVE alongside improved function and quality of life for this high-risk group, and ensuring that patients can continue to undertake exercise where it is not feasible to attend SEP, or where fluctuations in social-distancing restrictions occur.

Although TENS and behavioural interventions have been utilised previously in this population to improve physical activity. Neither MOSAIC or TENS have been utilised with aim to improve free living physical activity measured using an accelerometer, and there is a lack of data investigating these outcomes with home based exercise in general. While the author is aware of ongoing works investigating these outcomes, no trial to date has been developed a priori to evaluate the delivery of these treatments remotely in this population.

The primary aim of MAvERIC is to determine the acceptability and feasibility of electrical stimulation via a low-cost CE-marked device, and a remotely delivered walking based behavioural intervention (MOSAIC) in patients with PAD, compared to usual care.

The following research questions will be answered by this project:

1. What is the feasibility (i.e. recruitment and retention rates, adherence, safety, sample size for a definitive trial, potential for effectiveness) of conducting a definitive RCT utilising TENS or MOSAIC as an intervention compared to usual care?
2. How acceptable is TENS and MOSAIC interventions to patients with IC?
3. What are the effects of TENS and MOSAIC as interventions on free living physical activity, pain related, and quality of life PROMs?

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of symptomatic Peripheral Arterial Disease (PAD) including resting ABPI <0.9 in at least one leg
* Stable IC for ≥3 months
* Walking limited primarily by claudication
* Able to read and speak English to a level allowing satisfactory completion of the study procedures
* Able to provide written informed consent for participation

Exclusion Criteria:

* Planned surgical or endovascular intervention for PAD within the next 3 months
* Critical limb ischaemia
* The presence of any absolute contraindications to exercise testing/training as defined by the American College of Sports Medicine (ACSM)
* Previous experience of using TENS for PAD
* Contraindications to TENS (including epilepsy, dermatological conditions, indwelling electrical pumps/pacemakers) and inability to apply TENS independently.
* Patients who require walking aids including artificial limbs
* Major surgery, myocardial infarction or stroke/ TIA in the previous 6 months
* Co-morbidities that cause pain or limit walking to a greater extent than IC (e.g. severe arthritis, respiratory conditions)
* Severe peripheral neuropathies above the ankle.
* Participation in another research protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment rates | End of Study (12 weeks)
  Measure recruitment rates (ratio of patients who consent to participate to potentially eligible patient recorded via the study screening log
Participant retention rate | End of Study (12 weeks)
  Ratio of patients who completed the intervention and outcome assessment to the patient who consented
Adverse events | End of Study (12 weeks)
  Record defined adverse events in all groups
Uptake of interventions | End of Study (12 weeks)
  Measure uptake of intervention via log of TENS use and attendance at physiotherapy appointments and follow up phone calls
Qualitative analysis of participant experience of trial | End of Study (12 weeks)
  Analysis of semi-structured discussions with participants regarding experience of trial and interventions
Theoretical framework of acceptability (TFA) questionnaire | End of Study (12 weeks)
  Quantitative measurement of Acceptability of Intervention compared with usual care

SECONDARY OUTCOMES:
Change in daily physical activity | Baseline, 6 weeks, 12 weeks, 6 months (follow up), and 12 months (follow up)
  Total number of steps (activpal step counts)
Change in daily physical activity | Baseline, 6 weeks, 12 weeks, 6 months (follow up), and 12 months (follow up)
  Upright and sitting events
Change in daily physical activity | Baseline, 6 weeks, 12 weeks, 6 months (follow up), and 12 months (follow up)
  Walking events
Change in daily physical activity | Baseline, 6 weeks, 12 weeks, 6 months (follow up), and 12 months (follow up)
  Event-based claudication index (ratio of walking events to upright events) participants undertake in a day
Change in daily physical activity | Baseline, 6 weeks, 12 weeks, 6 months (follow up), and 12 months (follow up)
  Total duration of walking activity in minutes and seconds
Patient Reported Outcome Measure | Baseline, 6 weeks, 12 weeks, 6 months (follow up), and 12 months (follow up)
  Disease specific quality of life will be as assessed using the Intermittent Claudication Questionnaire (ICQ).
Patient Reported Outcome Measures | Baseline, 6 weeks, 12 weeks, 6 months (follow up), and 12 months (follow up)
  Generic quality of life via the EQ-5D-3L
Patient Reported Outcome Measures | Baseline, 6 weeks, 12 weeks, 6 months (follow up), and 12 months (follow up)
  Pain quality will be recorded using the Short Form McGill Pain Questionnaire (MPQ)
Patient Reported Outcome Measures | Baseline, 6 weeks, 12 weeks, 6 months (follow up), and 12 months (follow up)
  Average Pain intensity in the past 7 days will be recorded using a Visual Analogue Scale
Patient Reported Outcome Measures | Baseline, 6 weeks, 12 weeks, 6 months (follow up), and 12 months (follow up)
  Pain self-efficacy via. the Pain Self-Efficacy (PSEQ)
Patient Reported Outcome Measures | Baseline, 6 weeks, 12 weeks, 6 months (follow up), and 12 months (follow up)
  Pain Catastrophizing via. the Pain Catastrophizing Scale (PCS)

OTHER OUTCOMES:
Evaluation and monitoring of intervention fidelity | End of Study (12 weeks)
  This will be assessed by a member of the study team with reference to the MOSAIC materials and therapist training manual.

CONTACTS AND LOCATIONS:
Locations (1):
- NHS Lanarkshire, Glasgow, Lanarkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No